CLINICAL TRIAL: NCT05858489
Title: Concordance Between Mini-Mental Stats Examination (MMSE) and an Adapted Version of the MMSE in Reunion Island Population (MMS-Run) : Preliminary Study
Brief Title: Concordance Between Mini-Mental Stats Examination (MMSE) and an Adapted Version of the MMSE in Reunion Island Population (MMS-Run)
Acronym: MMS-R-ep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/30
Record Dates: First submitted 2023-04-25; First posted 2023-05-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Neurocognitive Deficit
Keywords: Neurocognitive Deficit; Neurocognitive Impairment; Major neurocognitive disorder; Dementia; Geriatric; Senior; Illeteracy : Mini Mental State Examination; Eldery
MeSH Terms: conditions — Dementia | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mini-Mental State Examination (MMSE) — Each patient will be evaluated by MMSE then by the adapted version of MMSE

SUMMARY:
Illeteracy concerns more than 38% of Réunion Island's people older than 65 years old, which makes it an important risk factor for dementia and a limit to neurocognitive test's administration.

The MMSRun is a Mini Mental State Examination's version adapted to illeteracy and Réunionese culture, inspired by Hindi Mental State Examination's work. It allows a way better participation during neurocognitive evaluation, but it has never been validated.

This study is a peliminary study to a validation, where the concordance between scores obtained from MMSRun and from the consensual version of Mini Mental State Examination proposed by GRECO (Groupe de Réflexion sur les Evaluations Cognitives) - the only french version validated - on a hospitalized and eldery population will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient who needs a cognitive evaluation by MMSe/MMS-RUN during usual medical care
* Patient born and living in Réunion Island
* Patient hospitalized in geriatrics department or in the departement of physical medecine and rehabilitation
* Patient who agrees to participate in the study and who does not oppose to the use of his data

Exclusion Criteria:

* Patient with hearing and visual disorder that can interfere in cognitive test administration
* Patient with altered state of consciousness (Glasgow score different of 15)
* Patient diagnosed or having symtoms compatible with a psychiatric pathology with psychosis (altered perception of reality)
* Patient with a current and severe addiction to Alcohol or any other drug (smoking excluded)
* Patient deprived of liberty by judicial or administrative decision and patient under curatorship or guardianship

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients will be selected in geriatric and physical medicine and rehabilitation departments at CHU de La Réunion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Total scoring of MMSE | Day 0
  30 questions, good response to a question = 1, bad response to a question = 0, global scoring between 0 and 30,
  Pathological threshold according to the socio-cultural level :
  * without diploma : total score <22
  * secondary education without the 3rd class : total score <23
  * secondary education from 3rd class to the senior year class (without bachelor degree)
  * higher education : total score <26
Total scoring of MMS-RUN | Day 1
  30 questions, good response to a question = 1, bad response to a question = 0, total score between 0 and 30,
  Pathological threshold according to the socio-cultural level :
  * without diploma : total score <22
  * secondary education without the 3rd class : total score <23
  * secondary education from 3rd class to the senior year class (without bachelor degree)
  * higher education : total score <26

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte CASALONGA, MD, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No